CLINICAL TRIAL: NCT04839978
Title: Community Randomized Trial in the Cherokee Nation: Connect and CMCA for Preventing Drug Misuse Among Older Adolescents
Brief Title: Community Trial in the Cherokee Nation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelli Komro, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000404; UH3DA050234 (NIH); UG3DA050234 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Opioid Abuse
Keywords: American Indian; Cherokee Nation; Community intervention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Sixteen to 20 high schools and surrounding towns within the 14 counties that partially or fully fall within the Cherokee Nation reservation in northeast Oklahoma will be randomly assigned to receive the preventive interventions offered by this study or usual school and community prevention. A total of 800 to 1200 students are expected to enroll from the randomized sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive Intervention (Experimental): Students in schools assigned to the preventive intervention study condition will take part in the Connect school-based prevention program and the community-level Communities Mobilizing for Change and Action (CMCA) intervention.
  Interventions: Behavioral: Connect Program; Behavioral: Communities Mobilizing for Change and Action (CMCA)
- Control Group (No Intervention): Students in schools assigned to the control group will not receive the Connect and CMCA interventions. Schools in the control group will receive usual school and community prevention and will be offered the trial's programs after the end of this three-year study.

INTERVENTIONS:
Behavioral: Connect Program — The Connect program includes school-based screening, brief intervention and referral, and will be treated as part of the participating schools' prevention programs. A computer-based screening and brief intervention will be supported by Cherokee Nation Behavioral Health (CNBH) supervised Connect coaches universally, to reduce potential stigma associated with speaking to a Connect coach and to reinforce drug free norms among all students. Follow-up of moderate to high-risk youth will be conducted by a Connect Coach through Zoom, other electronic communication, or in-person visits, with referral to Cherokee Nation or community services if deemed necessary.
  Arms: Preventive Intervention
Behavioral: Communities Mobilizing for Change and Action (CMCA) — The community-level intervention Communities Mobilizing for Change and Action (CMCA) will involve educating and organizing of adult volunteers and consent will be assumed by their participation. Trainings and tools will be provided, including Family Action Kits, to support local families, community organizations and citizens, including information on national and local opioid and other drug use, evidence-based policies, programs and practices, and how to motivate and create family and local action for drug prevention.
  Arms: Preventive Intervention

SUMMARY:
The target population is students attending high schools in small rural towns in the 14 counties that partially or fully fall within the Cherokee Nation reservation. Following recruitment of 20 school-based clusters, clusters are allocated to either the intervention condition or delayed-intervention control condition using constrained randomization. Constrained randomization helps to ensure balanced cluster sizes as well as similar levels of risk between the intervention and control at baseline. Study participants include all 10th grade students enrolled in the participating study high schools and students will be followed into the first year after their expected graduation.

DETAILED DESCRIPTION:
The national public health opioid crisis has disproportionately burdened rural White populations, and disproportionately burdened American Indian populations. Therefore, the Cherokee Nation (CN) and Emory University public health scientists have designed an opioid prevention trial to be conducted in at-risk rural communities in the CN (in northeast Oklahoma) with primarily White and American Indian adolescents and young adults. The goal of this study is to implement and evaluate a theory-based, integrated multi-level community intervention designed to prevent the onset and escalation of opioid and other drug misuse. The researchers propose a cluster randomized trial building directly on the success of their most recent previous trial, which demonstrated that the intervention effectively reduced alcohol and other drug use among American Indian and other youth living within the CN. Two distinct intervention approaches-community organizing as implemented in the established Communities Mobilizing for Change and Action (CMCA) intervention protocol, and universal school-based brief intervention and referral as implemented in the established Connect intervention protocol -will be expanded and integrated to further enhance effects in preventing and reducing opioid misuse. The CMCA and Connect interventions were originally designed to target adolescent alcohol use but nevertheless showed significant beneficial effects on use of other drugs, including prescription drug misuse. The proposed study will: (1) further improve the design of the interventions with increased focus on opioids, (2) test the expanded, integrated versions in a cluster randomized trial, and (3) design and test new systems for sustained implementation within existing structures of the Cherokee Nation. Building upon the extant prevention science evidence, this study will respond to a gap in evidence concerning opioid misuse prevention among at-risk adolescents transitioning to young adulthood among American Indian and other rural youth.

ELIGIBILITY:
Inclusion Criteria:

* Tenth grade students enrolled in the participating high schools

Exclusion Criteria:

* unable to understand written or verbal English

Inclusion criteria for high schools:

* Counties that partially or fully fall within the Cherokee Nation reservation
* Town population of 3,000 or less
* Class size between 30 to 100 students

Exclusion criteria for high schools:

* Metropolitan and micropolitan cores (Rural-Urban Commuting Area codes of 1 and 4)
* Existence of a community drug prevention coalition

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 919 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Komro, PhD, Principal Investigator — Emory University
Locations (1):
- Cherokee Nation Reservation, Tahlequah, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available for sharing, provided all data requests are reviewed and approved by the Cherokee Nation Institutional Review Board (IRB). Data and associated documentation sharing requires a negotiated data-sharing agreement that provides for: 1) review and approval of the data request and study protocol by the Cherokee Nation IRB, 2) a commitment to using the data only for research purposes, 3) restrictions against attempting to identify study participants, 4) a commitment to securing the data using secure computer technology, 5) a commitment to destroying data after the specific requested analyses are completed, 6) agreement to submit all presentations and manuscripts to the appropriate tribal authorities for review and approval prior to public dissemination and publication, 7) reporting responsibilities to the Cherokee Nation, 8) restrictions on redistribution of the data to third parties, and 9) proper acknowledgement of the source of the data.
Time Frame: Data will available for sharing following publication of the study findings.
Access Criteria: It is the responsibility of any external party requesting access to project data to request in writing to the project PI the specific data requested, and to apply to the Cherokee Nation IRB for such access according to procedures promulgated by the Cherokee Nation. Further, any such access is conditional on meeting all requirements specified by the Cherokee Nation IRB. Persons interested in using the data should contact the PI listed on manuscripts and publications as a means of facilitating access to the data.

REFERENCES:
- [Derived] Komro KA, Livingston MD, Skinner JR, Livingston BJ, Kominsky TK, Jagtiani A, Barry CM, Wagenaar AC, Cooper HLF, Harmon M, Ivanich E, LaBounty H, Gassaway AN, Talavera-Brown SL. Primary Prevention of Drug Overdoses in Rural Low-Resource and Tribal Communities: A Cluster Randomized Trial. Am J Public Health. 2025 Sep;115(9):1508-1517. doi: 10.2105/AJPH.2025.308205. PMID 40768695
- [Derived] Jagtiani A, Livingston MD, Barry CM, Talavera-Brown S, LaBounty H, Skinner JR, Livingston BJ, Lincoln AN, Komro KA. Tribal Identity, Pain Interference, and Substance Use Among American Indian and Alaska Native Adolescents. JAMA Pediatr. 2024 Nov 1;178(11):1192-1198. doi: 10.1001/jamapediatrics.2024.3284. PMID 39312248
- [Derived] Komro KA, Kominsky TK, Skinner JR, Livingston MD, Livingston BJ, Avance K, Lincoln AN, Barry CM, Walker AL, Pettigrew DW, Merlo LJ, Cooper HLF, Wagenaar AC. Study protocol for a cluster randomized trial of a school, family, and community intervention for preventing drug misuse among older adolescents in the Cherokee Nation. Trials. 2022 Feb 23;23(1):175. doi: 10.1186/s13063-022-06096-0. PMID 35197100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 919 participants were enrolled from 20 high schools in the Cherokee Nation Reservation, in Tahlequah, Oklahoma, USA. Participant enrollment began on September 29, 2021 (the day of the Baseline survey) and the assessment at the end of high school (spring of 12th grade) occurred on May 17, 2024. The final study assessment for the 6-months post-graduation time point occurred on December 31, 2024.
Units Other Than Participants: high schools
Groups:
- Preventive Intervention: Students in schools assigned to the preventive intervention study condition taking part in the Connect school-based prevention program and the community-level Communities Mobilizing for Change and Action (CMCA) intervention.
  The Connect program includes school-based screening, brief intervention and referral, and was treated as part of the participating schools' prevention programs. A computer-based screening and brief intervention was supported by Cherokee Nation Behavioral Health (CNBH) supervised Connect coaches universally, to reduce potential stigma associated with speaking to a Connect coach and to reinforce drug free norms among all students. Follow-up of moderate to high-risk youth was conducted by a Connect Coach through Zoom, other electronic communication, or in-person visits, with referral to Cherokee Nation or community services if deemed necessary.
  The community-level intervention Communities Mobilizing for Change and Action (CMCA) involved educating and organizing of adult volunteers and consent was assumed by their participation. Trainings and tools were provided, including Family Action Kits, to support local families, community organizations and citizens, including information on national and local opioid and other drug use, evidence-based policies, programs and practices, and how to motivate and create family and local action for drug prevention.
- Control Group: Students in schools assigned to the control group did not receive the Connect and CMCA interventions. Schools in the control group received usual school and community prevention and were offered the trial's programs after the end of this three-year study.
Period: Overall Study
Arm/Group | Preventive Intervention | Control Group
Started | 465; 10 high schools | 454; 10 high schools
Completed (Completed the Spring of 12th grade assessment.) | 330; 10 high schools | 307; 10 high schools
Not Completed | 135; 0 high schools | 147; 0 high schools
Not completed — Lost to Follow-up | 135 | 147

BASELINE CHARACTERISTICS:
Groups:
- Preventive Intervention: Students in schools assigned to the preventive intervention study condition taking part in the Connect school-based prevention program and the community-level Communities Mobilizing for Change and Action (CMCA) intervention.
- Total: Total of all reporting groups
Arm/Group | Preventive Intervention | Control Group | Total
Number analyzed (Participants) | 465 | 454 | 919
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (0.6) | 15.6 (0.7) | 15.5 (0.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 230 | 214 | 444
  Male | 215 | 222 | 437
  Decline to answer | 20 | 15 | 35
  Missing | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Only | 130 | 136 | 266
  White Only | 174 | 149 | 323
  American Indian and White | 102 | 103 | 205
  Other | 55 | 61 | 116
  Missing | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 465 | 454 | 919
Participants reporting alcohol use in past 30 days [Count of Participants; unit: Participants]
  Alcohol use reported | 74 | 92 | 166
  Missing response | 5 | 2 | 7
Participants reporting heavy alcohol use in past 30 days [Count of Participants; unit: Participants]
  Heavy alcohol use reported | 43 | 52 | 95
  Missing response | 4 | 7 | 11
Participants reporting marijuana use in past 30 days [Count of Participants; unit: Participants]
  Marijuana use reported | 68 | 68 | 136
  Missing response | 7 | 9 | 16
Participants reporting prescription opioid misuse in past 30 days [Count of Participants; unit: Participants]
  Prescription opioid misuse reported | 21 | 17 | 38
  Missing response | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Days of Alcohol Use
Description: The number of days of alcohol use in the past 30 days is compared between study arms.
Time Frame: Surveys were administered each fall and spring semester from baseline (fall of 10th grade) to spring of 12th grade (up to 31 months and 19 days)
Population: The analysis population includes participants who completed the baseline survey as the overall number of participants analyzed. The least squares means are calculated adjusting for repeated measures with responses from all participants in the baseline population. The number of participants at each time point represents the students who completed subsequent surveys at the indicated time points. Some survey items were left unanswered by students.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
days
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 425 | 414
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 0.71 (0.17) | 0.58 (0.14)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 384 | 372
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 0.70 (0.16) | 0.70 (0.16)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 364 | 341
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 0.69 (0.15) | 0.84 (0.18)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 334 | 322
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 0.68 (0.16) | 1.01 (0.22)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 324 | 305
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 0.66 (0.17) | 1.21 (0.28)

2. Primary Outcome: Number of Days of Heavy Alcohol Use
Description: The number of days of heavy alcohol use in the past 30 days is compared between study arms. Heavy alcohol use is defined as having at least four (among young women) or five (among young men) alcoholic drinks within a couple of hours.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
days
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 425 | 407
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 0.51 (0.11) | 0.30 (0.07)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 385 | 368
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 0.50 (0.10) | 0.40 (0.09)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 364 | 337
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 0.48 (0.10) | 0.52 (0.11)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 334 | 318
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 0.47 (0.10) | 0.68 (0.14)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 325 | 301
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 0.46 (0.11) | 0.90 (0.20)

3. Primary Outcome: Number of Days of Marijuana Use
Description: The number of days of marijuana use in the past 30 days is compared between study arms.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
days
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 418 | 402
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 1.53 (0.20) | 1.71 (0.22)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 381 | 367
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 1.50 (0.18) | 1.88 (0.21)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 360 | 330
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 1.46 (0.18) | 2.07 (0.23)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 328 | 316
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 1.44 (0.19) | 2.28 (0.27)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 322 | 298
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 1.41 (0.22) | 2.51 (0.35)

4. Primary Outcome: Number of Days of Opioid Misuse
Description: The number of days of opioid drug misuse use in the past 30 days is compared between study arms.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
days
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 414 | 392
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 0.24 (0.09) | 0.07 (0.04)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 376 | 357
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 0.19 (0.07) | 0.10 (0.04)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 350 | 320
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 0.15 (0.05) | 0.13 (0.05)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 323 | 307
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 0.12 (0.05) | 0.17 (0.07)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 319 | 293
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 0.10 (0.05) | 0.23 (0.10)

5. Secondary Outcome: Social Support From Parent/Caregiver
Description: Social support from parents/caregivers is assessed with 6 items which are responded to on a 4-point scale where 1 = never and 4 = often. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater support.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 422 | 409
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 3.50 (0.03) | 3.45 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 385 | 367
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 3.50 (0.03) | 3.47 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 356 | 341
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 3.49 (0.02) | 3.48 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 328 | 315
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 3.49 (0.03) | 3.50 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 323 | 301
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 3.49 (0.03) | 3.51 (0.03)

6. Secondary Outcome: Social Support From Friend
Description: Social support from a friend is assessed with 6 items, which are responded to on a 4-point scale where 1 = never and 4 = often. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater support.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 430 | 402
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 3.43 (0.03) | 3.39 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 392 | 365
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 3.43 (0.03) | 3.40 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 362 | 337
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 3.44 (0.03) | 3.41 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 329 | 312
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 3.44 (0.03) | 3.43 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 325 | 296
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 3.44 (0.04) | 3.44 (0.04)

7. Secondary Outcome: Social Support From Teacher
Description: Social support from a teacher is assessed with 6 items, which are responded to on a 4-point scale where 1 = never and 4 = often. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater support.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 419 | 399
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 3.25 (0.03) | 3.19 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 384 | 362
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 3.27 (0.03) | 3.22 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 355 | 332
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 3.29 (0.03) | 3.25 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 330 | 311
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 3.31 (0.03) | 3.28 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 316 | 296
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 3.33 (0.04) | 3.31 (0.04)

8. Secondary Outcome: Social Support From Other Adult
Description: Social support from an adult, other than a parent/caregiver or teacher, is assessed with 6 items which are responded to on a 4-point scale where 1 = never and 4 = often. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater support.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 427 | 407
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 3.05 (0.05) | 3.06 (0.05)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 386 | 365
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 3.09 (0.04) | 3.09 (0.04)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 362 | 334
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 3.14 (0.04) | 3.11 (0.04)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 332 | 310
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 3.18 (0.05) | 3.13 (0.05)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 322 | 293
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 3.22 (0.05) | 3.15 (0.05)

9. Secondary Outcome: Perceived Availability of Alcohol
Description: Ease or difficulty in accessing alcohol is assessed with 4 items using a 4-point scale where 1 = very difficult to get and 4 = very easy to get. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater ease of availability.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 422 | 404
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.18 (0.07) | 2.22 (0.07)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 386 | 366
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.20 (0.06) | 2.27 (0.07)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 360 | 337
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.22 (0.06) | 2.32 (0.07)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 331 | 311
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.24 (0.07) | 2.37 (0.07)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 324 | 295
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.26 (0.07) | 2.42 (0.07)

10. Secondary Outcome: Perceived Availability of Marijuana
Description: Ease or difficulty in accessing marijuana is assessed with 5 items using a 4-point scale where 1 = very difficult to get and 4 = very easy to get. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater ease of availability.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 418 | 403
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.04 (0.07) | 2.10 (0.07)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 387 | 362
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.06 (0.07) | 2.14 (0.07)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 360 | 335
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.08 (0.07) | 2.18 (0.07)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 331 | 309
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.10 (0.07) | 2.23 (0.07)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 322 | 296
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.12 (0.07) | 2.27 (0.07)

11. Secondary Outcome: Perceived Availability of Prescription Opioids
Description: Ease or difficulty in accessing prescription opioids is assessed with 5 items using a 4-point scale where 1 = very difficult to get and 4 = very easy to get. The total score is expressed as the mean across items and ranges from 1 to 4, with higher scores indicating greater ease of availability.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 422 | 404
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 1.52 (0.04) | 1.47 (0.04)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 389 | 359
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 1.51 (0.03) | 1.49 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 362 | 330
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 1.49 (0.03) | 1.51 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 335 | 312
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 1.48 (0.03) | 1.53 (0.04)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 326 | 294
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 1.47 (0.04) | 1.55 (0.04)

12. Secondary Outcome: Social Normative Beliefs About Alcohol Use
Description: Participants are asked 4 items to assess if they think various social groups (parents, community adults, peers, self) disapprove of young people drinking alcohol. Responses are given as 1 = don't disapprove, 2 = disapprove, and 3 = strongly disapprove. The total score is expressed as the mean across items and ranges from 1 to 3, with higher scores indicating stronger disapproval
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 423 | 399
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.11 (0.03) | 2.03 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 385 | 353
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.10 (0.03) | 2.02 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 357 | 332
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.10 (0.03) | 2.01 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 326 | 309
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.09 (0.03) | 2.00 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 325 | 291
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.08 (0.03) | 1.99 (0.03)

13. Secondary Outcome: Social Normative Beliefs About Marijuana
Description: Participants are asked 4 items to assess if they think various social groups (parents, community adults, peers, self) disapprove of young people using marijuana. Responses are given as 1 = don't disapprove, 2 = disapprove, and 3 = strongly disapprove. The total score is expressed as the mean across items and ranges from 1 to 3, with higher scores indicating stronger disapproval.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 423 | 396
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.16 (0.03) | 2.08 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 385 | 355
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.16 (0.03) | 2.09 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 353 | 331
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.16 (0.03) | 2.09 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 323 | 308
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.16 (0.03) | 2.09 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 319 | 292
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.15 (0.04) | 2.10 (0.04)

14. Secondary Outcome: Social Normative Beliefs About Prescription Opioids
Description: Participants are asked 4 items to assess if they think various social groups (parents, community adults, peers, self) disapprove of young people missing prescription opioids. Responses are given as 1 = don't disapprove, 2 = disapprove, and 3 = strongly disapprove. The total score is expressed as the mean across items and ranges from 1 to 3, with higher scores indicating stronger disapproval.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 424 | 400
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.54 (0.03) | 2.46 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 382 | 353
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.55 (0.02) | 2.49 (0.02)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 351 | 329
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.56 (0.02) | 2.51 (0.02)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 323 | 309
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.57 (0.03) | 2.54 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 319 | 292
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.58 (0.03) | 2.56 (0.03)

15. Secondary Outcome: Self-Efficacy
Description: Self-efficacy is assessed with 3 items asking how easy or hard it would be for participants to ask for help or refuse alcohol or drugs. Responses given on a 4-point scale, where 1 = very easy and 4 = very hard. The total score is expressed as the mean across items and ranges from 1 to 4, with lower scores indicating increased self-efficacy.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 428 | 413
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 1.59 (0.03) | 1.65 (0.03)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 388 | 372
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 1.58 (0.02) | 1.64 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 365 | 341
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 1.57 (0.02) | 1.63 (0.02)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 331 | 320
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 1.55 (0.03) | 1.62 (0.03)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 323 | 303
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 1.54 (0.04) | 1.60 (0.04)

16. Secondary Outcome: Normative Estimates of Peer Drug Use
Description: Normative estimates of peer drug use (alcohol, marijuana, prescription opioid misuse) are assessed with 3 items asking about how many of their peers in school used drugs in the past year. Possible responses are 1 = none or almost none, 2 = less than half, 3 = about half, 4 = more than half, and 5 = almost all or all. The total score is expressed as the mean across items and ranges from 1 to 5, with higher scores indicating higher normative estimates of peer drug use.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Intervention | Control Group
Number analyzed (Participants) | 465 | 454
score on a scale
  Baseline (Fall of 10th Grade) to Spring of 10th Grade: number analyzed (Participants) | 427 | 410
  Baseline (Fall of 10th Grade) to Spring of 10th Grade | 2.50 (0.06) | 2.51 (0.06)
  Baseline (Fall of 10th Grade) to Fall of 11th Grade: number analyzed (Participants) | 389 | 370
  Baseline (Fall of 10th Grade) to Fall of 11th Grade | 2.45 (0.06) | 2.52 (0.06)
  Baseline (Fall of 10th Grade) to Spring of 11th Grade: number analyzed (Participants) | 364 | 338
  Baseline (Fall of 10th Grade) to Spring of 11th Grade | 2.41 (0.06) | 2.52 (0.06)
  Baseline (Fall of 10th Grade) to Fall of 12th Grade: number analyzed (Participants) | 332 | 317
  Baseline (Fall of 10th Grade) to Fall of 12th Grade | 2.36 (0.06) | 2.52 (0.06)
  Baseline (Fall of 10th Grade) to Spring of 12th Grade: number analyzed (Participants) | 330 | 301
  Baseline (Fall of 10th Grade) to Spring of 12th Grade | 2.32 (0.07) | 2.52 (0.07)

17. Secondary Outcome: Number of Days of Alcohol Use
Description: The number of days of alcohol use in the past 30 days is compared between study arms.
Time Frame: 6 Months Post-Graduation
Reporting Status: Not Posted

18. Secondary Outcome: Number of Days of Heavy Alcohol Use
Description: as for outcome 2
Time Frame: 6 Months Post-Graduation
Reporting Status: Not Posted

19. Secondary Outcome: Number of Days of Marijuana Use
Description: The number of days of marijuana use in the past 30 days is compared between study arms.
Time Frame: 6 Months Post-Graduation
Reporting Status: Not Posted

20. Secondary Outcome: Number of Days of Opioid Drug Misuse
Description: The number of days of prescription opioid misuse in the past 30 days is compared between study arms.
Time Frame: 6 Months Post-Graduation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected on days when the surveys were administered, during the period of time of survey administration. Surveys were administered each fall and spring semester from baseline (fall of 10th grade) to spring of 12th grade and the final survey was administered at 6-months post-graduation (up to 39 months and 3 days).
Arm/Group | Preventive Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/465 | 0/454
Serious Adverse Events (participants affected / at risk) | 0/465 | 0/454
Other Adverse Events (participants affected / at risk) | 0/465 | 0/454

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04839978/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT04839978/ICF_000.pdf